CLINICAL TRIAL: NCT02880540
Title: The Use of Dexmedetomidine as an Adjuvant for Perioperative Pain Management in Morbidly Obese Adolescents Undergoing Bariatric Surgery
Brief Title: Dexmedetomidine to Treat Bariatric Surgery-associated Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janelle Vaughns (Other)
Responsible Party: Sponsor-Investigator, Janelle Vaughns, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00006562
Record Dates: First submitted 2016-05-12; First posted 2016-08-26 (Estimated); Results first posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Obesity
Keywords: Adolescent; Bariatric; Obesity; Pain; Opiate-sparing
MeSH Terms: conditions — Obesity; Pain | interventions — Fentanyl; Morphine; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): Fentanyl 50 micrograms IV every 15 minutes up to 3 doses in postanesthesia recovery room and Morphine 2mg IV every 2 hours for 2days on hospital floor
  Interventions: Drug: Fentanyl; Drug: Morphine
- Dexmedetomidine Treated (Experimental): Dexmedetomidine IV bolus 1.5microgram/kilogram and a continuous infusion starting at 0.1 microgram/kilogram/hour during surgery
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Fentanyl
  Other Names: Sublimaze
  Arms: Control Group
Drug: Morphine
  Arms: Control Group
Drug: Dexmedetomidine
  Arms: Dexmedetomidine Treated

SUMMARY:
Obesity represents one of the most important public health issues according to the World Health Organization and it has reached epidemic proportions globally. The prevalence of childhood obesity has rapidly increased over the past decade and is associated with multiple co-morbid disease states . It is estimated that approximately 15.5% of children and adolescents are obese with a body mass index of ≥95th percentile for age . This not only poses health concerns for the patient, but also places increased demands on our healthcare system that is already overwhelmed by burgeoning costs. Moreover, obese children and adolescents who maintain excessive weight as adults are predisposed to cardiovascular disease and premature death.

In carefully selected patients who have failed to lose weight by diet and exercise, bariatric surgery provides an option to obtaining a healthy weight.

It is increasingly becoming an attractive option, with the number of adolescents undergoing bariatric surgery in the United States tripling between 2000 and 2003.

Obese patients are often afflicted with multi-organ dysfunction and obstructive sleep apnea, which presents unique challenges to the anesthesiologist managing their perioperative care . Bariatric surgery in obese adolescents may be associated with significant postoperative pain. Potent intravenous opioids such as fentanyl and morphine are at the mainstay of perioperative pain management. Unfortunately, respiratory depression and airway obstruction can often occur following administration of opioids in obese patients . This makes providing a safe analgesic regimen difficult during the perioperative setting. As opioids can be associated with respiratory depression and upper airway obstruction, surgeons and anesthesiologists alike must reconcile the adequacy of pain control with the risk of respiratory complications after surgery in obese adolescents.

DETAILED DESCRIPTION:
Dexmedetomidine is a non-opioid drug that has shown some utility during bariatric surgery in the adult population because of its analgesic properties. It is a lipophilic imidazole derivative that is a selective α2-adrenoreceptor agonist with sedative and analgesic properties devoid of respiratory depressant effects . Dexmedetomidine produces sedation by modulating the release of the neurotransmitter norepinephrine within the locus coeruleus of the brain, which is vital to producing an awake state. In addition, by directly stimulating α2-receptors in the spinal cord, dexmedetomidine inhibits the firing of nociceptive neurons responsible for the propagation of pain signals.

Although dexmedetomidine is an agent with many off-label clinical applications in the pediatric setting, much about its pharmacokinetic and pharmacodynamics properties remain unknown. This is even more evident for pediatric patients that are obese. Currently, there are no reported pharmacokinetic and pharmacodynamic studies that have investigated dexmedetomidine in obese children and adolescents. Our previous experience with the use of dexmedetomidine in the perioperative period along with our robust obese surgical population certainly supports the notion that we are well poised to conduct the proposed trial

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 95th percentile.
* Hospitalized overnight after surgery

Exclusion Criteria:

* History or a family (parent or sibling) history of malignant hyperthermia
* Renal or hepatic disorders
* Allergy to opioid analgesics
* An allergy to α2-adrenergic agonists or sulfa drugs
* Uncontrolled hypertension
* Clinically significant neurologic diseases
* Pregnancy or lactating female

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2016-03; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Celeste Martin, MD, Principal Investigator — Childrens National Health System
Locations (1):
- Childrens National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Freedman DS, Mei Z, Srinivasan SR, Berenson GS, Dietz WH. Cardiovascular risk factors and excess adiposity among overweight children and adolescents: the Bogalusa Heart Study. J Pediatr. 2007 Jan;150(1):12-17.e2. doi: 10.1016/j.jpeds.2006.08.042. PMID 17188605
- [Background] Thompson DR, Obarzanek E, Franko DL, Barton BA, Morrison J, Biro FM, Daniels SR, Striegel-Moore RH. Childhood overweight and cardiovascular disease risk factors: the National Heart, Lung, and Blood Institute Growth and Health Study. J Pediatr. 2007 Jan;150(1):18-25. doi: 10.1016/j.jpeds.2006.09.039. PMID 17188606
- [Background] Finkelstein EA, Fiebelkorn IC, Wang G. National medical spending attributable to overweight and obesity: how much, and who's paying? Health Aff (Millwood). 2003 Jan-Jun;Suppl Web Exclusives:W3-219-26. doi: 10.1377/hlthaff.w3.219. PMID 14527256
- [Background] Ogden CL, Yanovski SZ, Carroll MD, Flegal KM. The epidemiology of obesity. Gastroenterology. 2007 May;132(6):2087-102. doi: 10.1053/j.gastro.2007.03.052. PMID 17498505
- [Background] Inge TH, Krebs NF, Garcia VF, Skelton JA, Guice KS, Strauss RS, Albanese CT, Brandt ML, Hammer LD, Harmon CM, Kane TD, Klish WJ, Oldham KT, Rudolph CD, Helmrath MA, Donovan E, Daniels SR. Bariatric surgery for severely overweight adolescents: concerns and recommendations. Pediatrics. 2004 Jul;114(1):217-23. doi: 10.1542/peds.114.1.217. PMID 15231931
- [Background] Tsai WS, Inge TH, Burd RS. Bariatric surgery in adolescents: recent national trends in use and in-hospital outcome. Arch Pediatr Adolesc Med. 2007 Mar;161(3):217-21. doi: 10.1001/archpedi.161.3.217. PMID 17339501
- [Background] Adams JP, Murphy PG. Obesity in anaesthesia and intensive care. Br J Anaesth. 2000 Jul;85(1):91-108. doi: 10.1093/bja/85.1.91. No abstract available. PMID 10927998
- [Background] Benumof JL. Obesity, sleep apnea, the airway and anesthesia. Curr Opin Anaesthesiol. 2004 Feb;17(1):21-30. doi: 10.1097/00001503-200402000-00005. PMID 17021525
- [Background] Ingrande J, Lemmens HJ. Dose adjustment of anaesthetics in the morbidly obese. Br J Anaesth. 2010 Dec;105 Suppl 1:i16-23. doi: 10.1093/bja/aeq312. PMID 21148651
- [Background] Feld JM, Hoffman WE, Stechert MM, Hoffman IW, Ananda RC. Fentanyl or dexmedetomidine combined with desflurane for bariatric surgery. J Clin Anesth. 2006 Feb;18(1):24-8. doi: 10.1016/j.jclinane.2005.05.009. PMID 16517328
- [Background] Tufanogullari B, White PF, Peixoto MP, Kianpour D, Lacour T, Griffin J, Skrivanek G, Macaluso A, Shah M, Provost DA. Dexmedetomidine infusion during laparoscopic bariatric surgery: the effect on recovery outcome variables. Anesth Analg. 2008 Jun;106(6):1741-8. doi: 10.1213/ane.0b013e318172c47c. PMID 18499604
- [Background] Mason KP, Lerman J. Review article: Dexmedetomidine in children: current knowledge and future applications. Anesth Analg. 2011 Nov;113(5):1129-42. doi: 10.1213/ANE.0b013e31822b8629. Epub 2011 Aug 4. PMID 21821507

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We identified 13 patients who had received dexmedetomidine intraoperatively during the course of laporoscopic sleeve gastrectomy.
Groups:
- Control Group: Fentanyl 50 micrograms IV every 15 minutes up to 3 doses in postanesthesia recovery room and Morphine 2mg IV every 2 hours for 2days on hospital floor
  Fentanyl
  Morphine
- Dexmedetomidine Treated: Dexmedetomidine IV bolus 1.5microgram/kilogram and a continuous infusion starting at 0.1 microgram/kilogram/hour during surgery
  Dexmedetomidine
Period: Overall Study
Arm/Group | Control Group | Dexmedetomidine Treated
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Dexmedetomidine Treated | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 13 | 26
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 16 [15 to 17.3] | 18 [17 to 18] | 17 [16 to 17.65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 0 | 7
  Not Hispanic or Latino | 6 | 12 | 18
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Pain Scores (Numerical Rating Scale 0-10) Using the Faces Pain Scale-Revised
Description: Average pain scores during the day of surgery using the FPS-R rates pain on a scale from 1-10, with 0 representing "no pain" and 10 "very much pain. Each level accompanies a facial expression, ranging from content to distress.
Time Frame: From surgery until discharge from the hospital, an average of 48 hours.
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Control Group | Dexmedetomidine Treated
Number analyzed (Participants) | 13 | 13
Units on a scale | 5 [4 to 6] | 3.4 [3 to 4.3]

ADVERSE EVENTS:
Time Frame: From surgery through hospital discharge, an average of 48 hours
Description: All patients received standard of care treatment arms
Arm/Group | Control Group | Dexmedetomidine Treated
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-17): https://cdn.clinicaltrials.gov/large-docs/40/NCT02880540/Prot_SAP_000.pdf